CLINICAL TRIAL: NCT04791189
Title: Survey on the Expectations of Adolescents With Juvenile Idiopathic Arthritis (JIA) Regarding Knowledge and Communication With Health Care Professionals in the Field of Sexual Health, and Their Parents' Views on the Subject.
Brief Title: Survey on the Expectations of Adolescents With Juvenile Idiopathic Arthritis (JIA) Regarding Knowledge and Communication With Health Care Professionals in the Field of Sexual Health, and Their Parents' Views on the Subject. (SNAPS-JIA)
Acronym: SNAPS-JIA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Societe Francaise de Rhumatologie (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 SAVEL
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; Sexual health; Patient education; Needs assessment
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with juvenile rheumatoid arthritis aged from 18 to 45 years: * Major male or female patient [18 to 45 years of age] with juvenile idiopathic arthritis reported before the age of 16.
  * - Able to understand and complete the questionnaire online (speaking and reading French, with an internet connection for completion via RedCap°). ¬
  * - Able to give informed consent to participate
  * - Involving one's parents in the survey is not a prerequisite for inclusion.
  Interventions: Other: questionnaire
- Parents of patients with juvenile rheumatoid arthritis aged from 18 to 45 years: Parents of adult patients with JIA
  * - Parents able to understand and complete the questionnaire online (speaking and reading French, having an internet connection for completion via Red Cap°).
  * - Able to give informed consent to participate
  * - The parents must have been in charge of the patient as a teenager.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire to survey the needs of adolescents with juvenile idiopathic arthritis and the views of their parents in the area of sexual health.

SUMMARY:
Sexual health is a legitimate area to explore in the care of these patients, as it has such an impact on quality of life. However, addressing sexual health in a situation of chronic disease confronts the double societal taboo of disease and sexuality. Health professionals are uncomfortable because they are not trained to talk about the subject, especially in the presence of parents and with a teenager they have watched grow up.

In this context, a needs survey among juvenile idiopathic arthritis (JIA) patients and the point of view of their parents in the field of sexual health seems necessary.

Main objective: To determine the expectations of adolescents (aged 10-19 years) with juvenile idiopathic arthritis regarding knowledge and communication with health care professionals in the field of sexual health.

DETAILED DESCRIPTION:
This study is non-interventional, multi-centre and does not change current practice.

It will begin with the construction in a multidisciplinary team of two "needs assessment" questionnaires, the first for adult patients who have suffered from JIA, the second for their parents.

They will be drawn up by three sexologists, two rheumatologists, a pediatrician, a nurse from UTEP, a biostatistician, a statistician specializing in questionnaire metrology, two patients with JIA, two parents of JIA patients, and the Director of the ANDAR patient association.

These "needs assessment" questionnaires, entirely anonymous, will be composed of closed, Likert scale or semi-open questions.

The questionnaires will be implemented under RedCap° for patient associations.

The material necessary for the study (invitation letter + "patients"/"parents"-information letters + paper questionnaires for both surveys + pre-stamped letters) will be in paper format for hospital centres. These centres will ensure the follow-up of the study.

The invitation to participate in the survey by mailing or newsletter or association website will be made by the heads of patient associations.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Patients with juvenile rheumatoid arthritis aged from 18 to 45 years
* - Major male or female patient [18 to 45 years of age] with juvenile idiopathic arthritis reported before the age of 16.
* - Able to understand and complete the questionnaire online (speaking and reading French, with an internet connection for completion via RedCap°). ¬
* - Able to give informed consent to participate
* - Involving one's parents in the survey is not a prerequisite for inclusion.

Parents :

* Parents of patients with juvenile rheumatoid arthritis aged from 18 to 45 years
* - Parents of adult patients with JIA
* - Parents able to understand and complete the questionnaire online (speaking and reading French, having an internet connection for completion via Red Cap°).
* - Able to give informed consent to participate
* - The parents must have been in charge of the patient as a teenager.

Exclusion Criteria:

* Persons opposing participation in the study. The study information letters will specify that participation is consent to participate in the study.
* Protected persons

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: - Patients with juvenile rheumatoid arthritis aged from 18 to 45 years, and their parents
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Responses of JIA patients to a questionnaire on their expectations during adolescence regarding knowledge and communication with health professionals in the field of sexual health ("patient needs assessment" questionnaire) . | Day 1
  Responses of JIA patients to a questionnaire on their expectations during adolescence regarding knowledge and communication with health professionals in the field of sexual health ("patient needs assessment" questionnaire)

SECONDARY OUTCOMES:
Responses of JIA patients to a questionnaire on their expectations during adolescence regarding knowledge and communication with health professionals in the field of sexual health ("patient needs assessment" questionnaire) | Day 1
  Responses of JIA patients to a questionnaire on their expectations during adolescence regarding knowledge and communication with health professionals in the field of sexual health ("patient needs assessment" questionnaire) .
Responses of parents of JIA patients to a questionnaire on their child's assumed expectations during adolescence regarding knowledge and communication with health professionals in the field of sexual health ("parent needs assessment" questionnaire). | Day 1
  Responses of parents of JIA patients to a questionnaire on their child's assumed expectations during adolescence regarding knowledge and communication with health professionals in the field of sexual health ("parent needs assessment" questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Carine SAVEL, Principal Investigator — CHU de Clermont-Ferrand
Locations (15):
- France (15):
  - CHU Bordeaux Pellegrin, Bordeau
  - AP-HP, Boulogne-Billancourt
  - Hôpital de La Cavale Blanche, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHUGA - Hôpital Sud, Échirolles
  - CHR Metz-Thionville, Metz
  - Association Nationale de Défense contre l'Arthrite Rhumatoïde, Montpellier
  - CHU de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - CHU de Nice Hopital Pasteur, Nice
  - Association KOURIR, Paris
  - APHP La Pitié Salpétrière, Paris
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU Toulouse, Toulouse
  - Association France Spondyloarthrite, Tulle

REFERENCES:
- [Derived] Savel C, Chausset A, Berland P, Guiguet-Auclair C, Cabane L, Fautrel B, Gaudin P, Guillot P, Hayem G, Lafarge D, Merlin E, Peziere N, Sordet C, Trope S, Tournadre A, Malochet S, Cohen JD. Survey of adolescents' needs and parents' views on sexual health in juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2023 Sep 5;21(1):95. doi: 10.1186/s12969-023-00884-x. PMID 37670340